CLINICAL TRIAL: NCT00270114
Title: Recombinant Human Erythropoietin (r-HuEPO) in Patients With Low Hematocrit Levels to Facilitate Presurgical Autologous Blood Donation in Patients Undergoing Orthopedic Surgery (An Open-label Dose Finding Study)
Brief Title: A Study of the Safety and Effectiveness of Epoetin Alfa in Facilitating Self-donation of Blood Before Surgery in Patients Who Are Undergoing Orthopedic Surgery and Who Have Low Hematocrit Levels (the Percent of Red Blood Cells in Whole Blood)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005914
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Blood Transfusion; Orthopedic Procedures
Keywords: Anemia; blood transfusion, autologous; epoetin alfa; epogen; erythropoietin; orthopedic procedures; orthopedic surgery
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of epoetin alfa and to determine whether epoetin alfa will facilitate self-donation of blood before surgery in patients who have anemia, (as indicated by low hematocrit levels, the percent of red blood cells in whole blood) and who will be undergoing orthopedic surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients undergoing major orthopedic surgery frequently require blood transfusions both during and after the operation. A large percentage of patients are not able to pre-deposit their own blood for transfusion. Additionally, when a patient is anemic, as determined by a low hematocrit level, the amount of blood collected from the patient may not be sufficient to satisfy the amount required for transfusion. Further, complications such as the transmission of infectious diseases are possible with transfusions from other donors. Agents that can facilitate self-donation and reduce the need for transfusions from others may improve the overall safety of surgery. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that is used to treat anemia by stimulating red blood cell production. This is a randomized, open-label, placebo-controlled, parallel group, multicenter study to evaluate the safety of epoetin alfa and to determine whether epoetin alfa will facilitate the self-deposit of blood by patients who have low hematocrit levels, are undergoing orthopedic total hip replacement surgery, and are expected to require 3 to 4 units of blood during and after surgery. The study consists of a 5-day screening period when patients' study eligibility is determined, a 21-day treatment and blood collection period, and a period around the time of surgery (that includes recording the patient's blood status before surgery, as well as recording of blood loss and number of self-donated and/or donor-donated units of blood used during or after surgery). Eligible patients will be randomly assigned to one of four treatment groups: epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 600 U/kg, placebo to match the volume of epoetin alfa 300 U/kg, or placebo to match the volume of epoetin alfa 600 U/kg, by injection into a vein. Twice as many patients will receive epoetin alfa as will receive placebo. Patients and the physician will know the group to which an individual patient is assigned. Study medication will be administered to each patient every 3 to 4 days, for a total of 6 doses during the 21-day treatment period ending just before surgery. Additionally, all patients will receive 300 milligrams of an iron supplement daily by mouth or by a combination of an iron supplement by mouth and injected into a vein during the 21-day treatment period. The dose of the iron supplement and need for administration of an iron supplement into a vein will be determined based on a blood test measuring the iron content in the blood after each collection of blood for self-donation. Patients who are borderline iron-deficient at screening may be given iron injected into a vein 3 to 4 days before the start of the study. Thereafter, patients will be randomly assigned to receive either a daily oral iron supplement only or both a daily oral iron supplement plus iron injected into a vein after each collection of a unit of blood. On Day 1, before the first dose of study drug is given, one unit of blood will be collected and stored for self-donated blood transfusion during or after surgery, only from those patients whose red blood cell level shows they are not anemic, as determined by a hematocrit level >=35%. Every 3 to 4 days thereafter, the patients' blood will be analyzed and one unit of blood will be collected from each patient whose red blood cell level is >=35%. A maximum of 6 units of blood can be collected during the 3-week period before surgery and stored for self-donation. If sufficient units for surgery are not collected from a patient, preparations will be made for that patient to receive needed units of blood from donors. Safety evaluations will include laboratory tests, physical examination, vital signs, and recording of adverse events. The effectiveness of epoetin alfa will be evaluated by comparing the number of self-donated units of blood collected from each treatment group, the change in hemoglobin, the change in hematocrit (the percent of red blood cells in whole blood), and the number of immature red blood cells from before the start of the study to the end of the study. The study hypothesis is that treatment with epoetin alfa will facilitate self-donation of blood in patients with low hemoglobin and hematocrit levels who are undergoing orthopedic surgery. Epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 600 U/kg, or placebo, by injection into a vein; dose given twice weekly starting 3 weeks before surgery and ending just before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for hip replacement surgery
* having an anticipated requirement of 3 or more units of blood
* having a hematocrit level <=0.39
* having a hemoglobin level <= 12.5 grams/deciliter
* having laboratory tests within normal ranges, including stool negative for occult blood

Exclusion Criteria:

* Patients with a history of any blood disease
* having signs and symptoms of significant disease/dysfunction, or signs and symptoms of significant ongoing blood loss
* having uncontrolled high blood pressure, or a folate, vitamin B12, or iron deficiency, or signs and symptoms suggestive of an autoimmune disease causing blood to break down and release iron-containing pigment
* taking medication known to suppress the formation of red blood cells within 1 month before the start of the study
* having a history of seizures, or the presence of active inflammatory disease (e.g., rheumatoid arthritis), however, patients with osteoarthritis may be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Study Completion 1991-03 (Actual)

PRIMARY OUTCOMES:
Number of self-donated units of blood and the total volume of red blood cells donated; Number of blood units from other donors used for transfusion during surgery

SECONDARY OUTCOMES:
Changes in hemoglobin, hematocrit, red blood cell count, and effects of oral iron versus oral plus intravenous iron from before the study to the end of study; Assessment laboratory tests, vital signs, physical examination, and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of epoetin alfa in facilitating self-donation of blood before surgery in patients who are undergoing orthopedic surgery and who have low hematocrit levels (the percent of red blood cells in whole blood) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=683&filename=CR005914_CSR.pdf